CLINICAL TRIAL: NCT00191711
Title: Phase II Study of 6 Weeks Intravesical Gemcitabine Instillation Followed By Transurethral Resection in Patients Affected By Superficial Bladder Cancer at Low Risk
Brief Title: Intravesical Gemcitabine Instillation Followed by Transurethral Resection for the Treatment of Patients With Superficial Bladder Cancer at Low Risk.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8332; B9E-MC-S346
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Superficial Bladder Cancer
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — Gemcitabine

INTERVENTIONS:
Drug: Gemcitabine

SUMMARY:
The purpose of this study is to determine whether neoadjuvant intravesical Gemcitabine is enough active in patients with a solitary, low risk superficial bladder cancer.After diagnostic urethrocystoscopy or bladder sonography, all patients will receive intravesical gemcitabine once a week during 6 weeks. Two weeks after finishing antiblastic therapy, all patients will be submitted to a new cystoscopy, with TUR or cold biopsies of the site of the initial lesion.

ELIGIBILITY:
Inclusion Criteria:

* Primary solitary bladder tumour not exceeding 2 cm of diameter at sonography and/or at cystoscopy, judged by the investigator not muscle infiltrating and at low risk
* Urinary cytology negative for severe dysplasia (G3).
* ECOG performance status 0-1
* Absence of anti-coagulant therapy or acetyl-salicylic acid chronic therapy
* Absence of other present or past neoplasias except for healed skin basalioma

Exclusion Criteria:

* Tumours with infiltrative patterns at cystoscopy
* Transitional carcinoma of the upper urinary tract and prostatic urethra.
* Any previous or concomitant malignancy other than superficial bladder cancer with the exception of cutaneous basalioma and/or cancer of the cervix, adequately treated.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43
Dates: Start 2004-02; Study Completion 2005-10

PRIMARY OUTCOMES:
To evaluate pathological complete response rate achieved by 6 week neoadjuvant intravesical administration of Gemcitabine followed by transurethral resection (TUR) or cold biopsies, in patients affected by low risk superficial bladder cancer .

SECONDARY OUTCOMES:
To assess toxicity profile in the same group of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Monday-Friday 9 am-5 pm Eastern time (UTC/GMT - 5 hours, EST), Study Chair — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, please call 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559), Mon - Fri 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your physician, Sesto Fiorentino, Florence, Italy